CLINICAL TRIAL: NCT01208155
Title: An Open-label, Randomized, Four-way Crossover Study in Healthy Male Subjects to Assess the Relative Bioavailability of 4 Different Fostamatinib Tablets
Brief Title: Study in Healthy Males to Assess Bioavailability of 4 Different Fostamatinib Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00016
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Bioavailability; Pharmacokinetics
Keywords: Phase 1; Healthy; pharmacokinetics; Fostamatinib
MeSH Terms: interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Fostamatinib 50 mg tablet x 2
  Interventions: Drug: Fostamatinib
- 2 (Experimental): Fostamatinib 100 mg tablet (batch 1)
  Interventions: Drug: Fostamatinib
- 3 (Experimental): Fostamatinib 100 mg tablet (batch 2)
  Interventions: Drug: Fostamatinib
- 4 (Experimental): Fostamatinib 100 mg tablet (batch 4)
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Oral tablets, 50 mg x 2, single dose
  Arms: 1
Drug: Fostamatinib — Oral tablets, 100 mg Batch 1, single dose
  Arms: 2
Drug: Fostamatinib — Oral tablets, 100 mg Batch 2, single dose
  Arms: 3
Drug: Fostamatinib — Oral tablets, 100 mg Batch 3, single dose
  Arms: 4

SUMMARY:
Study in healthy males to assess bioavailability of 4 different fostamatinib tablets

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 50 kg and body mass index (BMI) between 18.0 and 35.0 kg/m2 inclusive
* Volunteers must be willing to use barrier contraception ie, condoms, from the Day 1 of Treatment Period 1 until 2 weeks after the final dosing of the investigational product (IP)

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs (except for cholecystectomy)
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of drug
* Volunteers who smoke more than 5 cigarettes or the equivalent in tobacco per day
* Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis results as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability of R406 when fostamatinib is administered as 50 mg tablets versus 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 1 until 96 hours post dose of each treatment period
Relative bioavailability of R406 when fostamatinib is administered as 50 mg tablets versus 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 2 until 96 hours post dose of each treatment period
Relative bioavailability of R406 when fostamatinib is administered as 50 mg tablets versus 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 3 until 96 hours post dose of each treatment period
Relative bioavailability of R406 when fostamatinib is administered as 50 mg tablets versus 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 4 until 96 hours post dose of each treatment period
Relative bioavailability of R406 when fostamatinib is administered as 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 1 until 96 hours post dose of each treatment period
Relative bioavailability of R406 when fostamatinib is administered as 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 2 until 96 hours post dose of each treatment period
Relative bioavailability of R406 when fostamatinib is administered as 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 3 until 96 hours post dose of each treatment period
Relative bioavailability of R406 when fostamatinib is administered as 3 different 100 mg tablet batches (assessment will include but is not limited to: plasma R406 AUC, Cmax ) | Daily during Treatment Period 4 until 96 hours post dose of each treatment period

SECONDARY OUTCOMES:
To examine the safety and tolerability of fostamatinib 50 mg and 100 mg tablet batches The safety endpoints will include: adverse event monitoring, vital signs, physical examinations, clinical laboratory tests, ECGs. | Screening, throughout the 4 treatment periods, and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, Study Director — AstraZeneca; Carlos Prendes, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States